CLINICAL TRIAL: NCT06008834
Title: First-day Discharge Enhanced Recovery After Surgery Protocol for Minimal Invasive Colorectal Surgery: Pilot Study
Brief Title: First-day Discharge Enhanced Recovery After Surgery Protocol for Minimal Invasive Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Anna Pallisera-Lloveras, MD, PhD, Corporacion Parc Tauli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIR2022020
Record Dates: First submitted 2023-08-23; First posted 2023-08-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Disorders; Surgery

STUDY DESIGN:
Intervention Model Description: Single Group Interventional Pilot Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Patients who undergo a minimal invasive colorectal surgery and are included in the first-day discharge protocol with domiciliary follow-up
  Interventions: Procedure: First-day discharge protocol

INTERVENTIONS:
Procedure: First-day discharge protocol — Enhance Recovery after Surgery (ERAS) protocol consisting in perioperative mesures and first-day hospital discharge with domiciliary follow-up

SUMMARY:
The enhanced recovery after surgery (ERAS) protocols are multimodal perioperative care pathways designed to achieve early recovery after surgical procedures by maintaining preoperative organ function and reducing the profound stress response following surgery. This type of approach has led to an earlier hospital discharge of patients with a low rate of postoperative complications.

Purpose: the aim of this study is to evaluate an ERAS protocol with fist-day hospital discharge and domiciliary follow-up for minimal invasive colectomy.

Method: unicenter pilot study of patients with indication of minimally invasive right colectomy or sigmidectomy who will follow an ERAS protocol according to international guidelines and will be discharged the first day of surgery with a domiciliary follow-up. Hospital readmission is considered as the primary outcome. A total sample of 40 cases is considered, with 20 right colectomies and 20 sigmoidectomies. An independent analysis of both techniques will be performed.

DETAILED DESCRIPTION:
Introduction: the enhanced recovery after surgery (ERAS) protocols are multimodal perioperative care pathways designed to achieve early recovery after surgical procedures by maintaining preoperative organ function and reducing the profound stress response following surgery. The key elements of ERAS protocols include preoperative counselling, optimization of nutrition, standardized analgesic and anesthetic regimens and early mobilization. This type of approach has led to an earlier hospital discharge of patients with a low rate of postoperative complications.

Purpose: the aim of this study is to evaluate an ERAS protocol with fist-day hospital discharge and domiciliary follow-up for minimal invasive colectomy.

Method: unicenter pilot study of patients with indication of minimally invasive right colectomy or sigmidectomy who will follow an ERAS protocol according to international guidelines and will be discharged the first day of surgery with a domiciliary follow-up.

Outcomes:

* Primary: hospital readmission
* Secondary: postoperative complications (Clavien-Dindo), domiciliary follow-up mean time before final postoperative discharge, emergency department re-consulting.

Sample: a total sample of 40 cases is considered, with 20 right colectomies and 20 sigmoidectomies.

Analysis: an independent analysis of both techniques will be performed. Pilot study without control branch.

ELIGIBILITY:
Inclusion Criteria:

* Pacients who undergo a minimal invasive sigmoidectomy or right colectomy.
* Benign or malignant desease.
* No expected stoma
* ASA ≤ III
* Family support

Exclusion Criteria:

* Emergency surgery
* Anticoagulant therapy
* Recent immunosupresor therapy (less than one month)
* Anemia (Male Hb >120 g/L, Female Hb >110 g/L)
* Malnutrition (Albumine >35 g/L)
* Dementia
* Moderate or high frailty
* Syncronic neoplasia
* Previous colorectal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Readmission | 30 days after surgery
  Hospital readmission after first-day hospital discharge

SECONDARY OUTCOMES:
Postoperative complications | 30 days after surgery
  Postoperative complications after first-day hospital discharge acording to Clavien-Dindo classification
Emergency Department re-consultation | 30 days after surgery
  Emergency Department re-consultation with no readmission after first-day hospital discharge
Domiciliary Follow-up | 30 days after surgery
  Domiciliary follow-up mean time before domiciliary discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pallisera-Lloveras, MD, PhD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital; Laura Mora-Lopez, MD, PhD, Study Director — Corporacio Parc Tauli. Parc Tauli University Hospital; Oriol Pino-Perez, MD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital
Locations (1):
- Parc Tauli University Hospital, Sabadell, Barcelona, Spain